CLINICAL TRIAL: NCT05551000
Title: Effects of Functional and Traditional Groups Class Training on Function and Health Among Female Older Adults: A Cluster-Randomized Controlled Trial
Brief Title: Functional vs Traditional Training in Older Women's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Lasse Engberg Treu Lassen, Ph.D. candidate, Aalborg University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 438956
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Performance Enhancement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): This group will use a functional training system developed specifically for elderlies to improve everyday movements, physical strength and balance.
  Interventions: Other: Experimental, comparator and control
- Positive control (Active Comparator): This group will use a general training system developed for elderlies to improve everyday movements, physical strength and balance.
  Interventions: Other: Experimental, comparator and control
- Negative control (No Intervention): Control group: A group that is not treated.

INTERVENTIONS:
Other: Experimental, comparator and control — To quantify the effect of a training intervention for elderlies on improved range of motion, dynamic balance, gait speed, gait coordination, everyday movements and strength compared to a training group from the Norwegian elderly concept "Stærk og Stødig" and a control group.
  Arms: Intervention; Positive control

SUMMARY:
This study investigates how balance, mobility, strength, gait speed, and health-related quality of life in older adults (65+) are affected after an 8-week training period using the Norwegian national concept for older adults, Strong and Steady, compared to a modified version that incorporates functional training variables.

ELIGIBILITY:
Inclusion Criteria:

* Elderlies aged 65 to 75 years old.
* Have been participating and physical training for at least six months before the start of the intervention.
* The participants must be highly motivated for the project, which will be measured using the likard scale.

Exclusion Criteria:

* Illness or injury within the last three months.
* Do not have the ability to complete the test battery concerning set minimum criteria

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Mobility test | Day 1
  Chair-sit-and-reach and back scratch test (Cm)
Mobility test | 2 months
  Chair-sit-and-reach and back scratch test (Cm)
Y-Balance Test | Day 1
  Measure balance performance (Cm)
Y-Balance Test | 2 months
  Measure balance performance (Cm)
Strength Test | Day 1
  Chair stand and Arm curl test (Repetitions)
Functional Strength Test | 2 months
  Chair stand and Arm curl test (Repetitions)
Time up-and-go test | Day 1
  Measure agility (Secounds)
Time up-and-go test | 2 months
  Measure agility (Secounds)
6-minute walking test | Day 1
  Measure walking distance (Meters)
6-minute walking test | 2 months
  Measure walking distance (Meters)
SF-36 questionnaire | 1 day
  Measure the participant's Health-related quality of life

SECONDARY OUTCOMES:
SF-36 questionnaire | 2 months
  Measure the participant's Health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- SSA Steinkjer, Steinkjer, Norway

IPD SHARING:
Plan to Share IPD: No